CLINICAL TRIAL: NCT06488209
Title: A Phase 1 Randomized, 3-Part, Placebo-Controlled, Single Ascending and Multiple Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of LAD191 in Healthy Subjects and Subjects With an Autoimmune Disease
Brief Title: Single and Multiple Ascending Dose Study in Healthy Participants and Participants With an Autoimmune Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: M-27134-01
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Parts 1 and 2 of the study will be single-blind and Part 3 will be double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part 1: LAD191 (Cohort 1) (Experimental): Participants will receive single ascending dose of LAD191 subcutaneous (SC) injection on Day 1.
  Interventions: Drug: LAD191
- Part 1: LAD191 (Cohort 2) (Experimental): Participants will receive single ascending dose of LAD191 SC injection on Day 1.
  Interventions: Drug: LAD191
- Part 1: LAD191 (Cohort 3) (Experimental): Participants will receive single ascending dose of LAD191 SC injection on Day 1.
  Interventions: Drug: LAD191
- Part 1: LAD191 (Cohort 4) (Experimental): Participants will receive single ascending dose of LAD191 SC injection on Day 1.
  Interventions: Drug: LAD191
- Part 1: LAD191 (Cohort 5) (Experimental): Participants will receive single ascending dose of LAD191 SC injection on Day 1.
  Interventions: Drug: LAD191
- Part 1: Placebo (Placebo Comparator): Participants will receive single dose of matching placebo SC injection on Day 1 (Cohort 1 to Cohort 5).
  Interventions: Other: Placebo
- Part 2: LAD191 (Cohort 6) (Experimental): Participants will receive multiple ascending doses of LAD191 SC injection on Days 1, 8, 15, 22, 29 and 36.
  Interventions: Drug: LAD191
- Part 2: LAD191 (Cohort 7) (Experimental): Participants will receive multiple ascending doses of LAD191 SC injection on Days 1, 8, 15, 22, 29 and 36.
  Interventions: Drug: LAD191
- Part 2: LAD191 (Cohort 8) (Experimental): Participants will receive multiple ascending doses of LAD191 SC injection on Days 1, 8, 15, 22, 29 and 36.
  Interventions: Drug: LAD191
- Part 2: Placebo (Placebo Comparator): Participants will receive multiple doses of matching placebo SC injection on Days 1, 8, 15, 22, 29 and 36 (Cohort 6 to Cohort 8).
  Interventions: Other: Placebo
- Part 3: LAD191 (Cohort 9) (Experimental): Participants will receive repeat doses of LAD191 SC injection on Days 1, 8, 15, 22, 29 and 36.
  Interventions: Drug: LAD191
- Part 3: Placebo (Placebo Comparator): Participants will receive repeat doses of matching placebo SC injection on Days 1, 8, 15, 22, 29 and 36 (Cohort 9).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LAD191 — LAD191 SC injection.
  Arms: Part 1: LAD191 (Cohort 1); Part 1: LAD191 (Cohort 2); Part 1: LAD191 (Cohort 3); Part 1: LAD191 (Cohort 4); Part 1: LAD191 (Cohort 5); Part 2: LAD191 (Cohort 6); Part 2: LAD191 (Cohort 7); Part 2: LAD191 (Cohort 8); Part 3: LAD191 (Cohort 9)
Other: Placebo — Matching placebo SC injection.
  Arms: Part 1: Placebo; Part 2: Placebo; Part 3: Placebo

SUMMARY:
The main purpose of this study is to to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity of LAD191 in healthy adults and in adults with an autoimmune disease.

DETAILED DESCRIPTION:
This is a 3-part study. Part 1 will be comprised of up to 5 cohorts of healthy adult participants and will investigate single ascending doses of LAD191. Part 2 will be comprised of up to 3 cohorts of healthy adult participants and will investigate multiple ascending doses of LAD191. Part 3 will be comprised of single cohort of participants with an autoimmune disease and will investigate repeat doses of LAD191. Each ascending dose level will be investigated by a sequential cohort, with dose escalation based on satisfactory safety, tolerability, PK, PD, immunogenicity, biomarker and clinical response assessments will be performed throughout.

Each cohort will be randomized to receive LAD191 and placebo.

Each participant will participate for about 14 weeks in Part 1, 17 weeks in Part 2 and 18 weeks in Part 3 of the study.

ELIGIBILITY:
Inclusion Criteria:

(Applicable to Both Healthy and an Autoimmune Disease Participants Unless Indicated Otherwise)

1. Participant provides written informed consent prior to any protocol related procedures, including screening evaluations. Participant must be able to understand the consent form and instructions and to provide consent directly; no guardian/legal representative or caregiver may provide consent for the participant.
2. Male or female, greater than or equal to (>=)18 and less than or equal to (<=) 65 years of age, with a body mass index (BMI) within the range of 18.5 to 29.9 kilogram per square meter (kg/m^2) (inclusive) and body weight of >=50 kilograms (kg).
3. Participant is healthy, in the clinical judgement of the Investigator, based medical history, physical examination, vital signs, ECG, and laboratory investigations (i.e., has clinical laboratory tests that are within the reference ranges or are clinically acceptable per Investigator judgment).
4. Participant has a seated systolic blood pressure (SBP) >=90 mm Hg and <=140 mm Hg or a seated diastolic BP (DBP) >=50 mm Hg or <=90 mm Hg.
5. Participant is willing and able to understand and comply with all aspects of the protocol.
6. Participant must agree to the following requirements during the study:

   * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result within 7 days prior to first dosing plus a negative urine pregnancy test pre-dose on Day 1 and must be willing to use a highly effective form of contraception (ICH E8 Guideline, 1997; (ICH M3 [R2] Guidance, 2009; (FDA M3 [R2] Guidance, 2010) for the duration of the study and for at least 3 months after the last dose of study medication. Methods like periodic abstinence, post-ovulation procedures and withdrawal are not considered adequate.
   * Males with partners of childbearing potential must be willing to use condoms in combination with a second effective method of contraception during the study. Male participants must continue to use contraception (condoms plus a second effective method) for 165 days following administration of the study drug.
   * Male participants must agree not to donate sperm during the study and for 165 days following administration of the study drug.

Participants with an Autoimmune Disease (Cohort 9 Only):

For participants with an autoimmune disease, the inclusion criteria for healthy participants listed above apply, with the following changes/additions:

1. Male or female, >=18 to <=65 years of age, with a BMI within the range 18.5 to 34.9 kg/ m^2, and body weight of >=50 kg.
2. Current diagnosis of an autoimmune disease by the Investigator and with signs and symptoms consistent with an autoimmune disease for at least 3 months prior to Day -1 (baseline).

Exclusion Criteria:

(Applicable to Both Healthy and an Autoimmune Disease Participants Unless Indicated Otherwise)

1. Participant has received treatment with LAD191 previously.
2. Known hypersensitivity to LAD191 or any of its excipients.
3. Hypersensitivity or reaction to a prior biologic (antibody-based) therapy (regardless of indication), that was clinically significant, as per judgment of Investigator.
4. History of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, inflammatory, or allergic disease (including drug allergies, any active seizure disorder requiring therapy with antiepileptic drugs, active peptic ulcer disease, gastrointestinal bleeding, chronic gastritis, inflammatory bowel disease or chronic diarrhea, but excluding mild seasonal allergies or stable, well-controlled thyroiditis). Note that participants with thyroid hormone deficiency, hypertension, hyperlipidemia, or diabetes mellitus may be included in Part 3 of the study.
5. Active chronic or acute infection requiring treatment with systemic antimicrobials, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Day -1, or superficial skin infections within 4 weeks prior to Day -1, or fever > 38°C during within 1 week before Day -1.
6. A positive test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) on Day -1, or the second negative test after a previous SARS CoV-2 infection was <=14 days before Day -1, or the participant's SARS CoV-2-associated symptoms resolved <=14 days before Day -1.
7. Presence of skin comorbidities that may interfere with study assessments, in the opinion of the Investigator.
8. Participant has current tuberculosis (TB) or any history of active or latent TB, regardless of prior treatment.
9. History of malignancy, regardless of outcome.
10. Participant has any condition that, in the opinion of the Investigator, would interfere with the PK evaluation of LAD191 or participant safety or the interpretation of study results
11. Clinically significant ECG abnormality, including, but not limited to, the following:

    * An abnormal PR interval (>=220 msec or <=100 msec).
    * QTc prolongation (corrected QT interval by Fredericia's formula [QTcF] >=450 msec).
    * Mean heart rate <=45 bpm or >100 bpm.
12. Known history of liver disease or clinically significant abnormal (as per judgment of Investigator) liver function test(s) at Screening (ALT, AST, alkaline phosphatase [ALP], or TBili >1.5 x ULN).
13. Impaired renal function (laboratory values out of the normal range that are clinically significant, as judged by the Investigator).
14. Congenital or acquired immunosuppressive condition that would put participant at risk during the study, per Investigator judgment.
15. Neutropenia; defined as a neutrophil count <2.0 x 10^9/L, at Screening.
16. Participant has had major surgery (requiring general anesthesia) within 3 months prior to Day -1, or has major surgery planned during the study. For participants with an autoimmune disease may have had incision and drainage of abscesses up to 1 week before Day -1).
17. Participant has donated plasma or blood or has lost more than 450 ml blood in the 60 days prior to Day -1, or intends to donate blood during the study or in the 60 days after the last scheduled study visit.
18. Participant is pregnant or breastfeeding (or is planning to become pregnant or breastfeed during the study or within 90 days after the last dose of study drug).
19. History of, or positive test result at Screening for, hepatitis B surface antigen (HBsAg), antibody to hepatitis B core antigen (anti-HBcAg), antibody to the hepatitis C virus (anti-HCV), or antibody to the human immunodeficiency virus (HIV-1/2).
20. Participant has taken any medications, including over-the-counter (OTC) medications, within 14 days (or at least 5 half-lives, whichever is longer) before Day -1. (Note that hormonal contraceptives are allowed, and acetaminophen is permitted at doses <=2 g/day up to 48 hours prior to each study visit).
21. Participant has received any type of live or attenuated vaccinations within 28 days prior to Screening, or is planning to receive any such vaccine during the study (inactive vaccines are allowed) or has received a SARS-CoV-2 vaccine within 14 days of Day 1.
22. Participant has received any investigational drug in any clinical study within 30 days (or at least 5 half-lives, whichever is longer) prior to Day -1, or is on extended follow-up from such a clinical study.
23. Participant has a history (within 2 years prior to Screening) of alcohol or drug abuse, as per Investigator judgment, or has a positive urine screen for drugs of abuse (opiates, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, cotinine, phencyclidine) at Screening or on Day -1, or a positive urine alcohol test at Screening or on Day -1.
24. Consumption of alcohol within 48 hours (2 days) before Day -1.
25. Participant is involved in strenuous physical activity or contact sports within 96 hours (4 days) prior to Day -1.
26. Consumption of any foods containing poppy seeds within 48 hours (2 days) prior to Screening and Day -1 as this could result in a false positive drug screen result.
27. Participant has any other serious or uncontrolled physical or mental dysfunction that, as judged by the Investigator, could place the participant at higher risk derived from his/her participation in the trial, could confound the results of the trial or is likely to prevent the participant from complying with the requirements of the trial or completing the trial.
28. Participant is an employee or relative of the Sponsor/vendors, clinical study site, or is an individual or employee directly involved with the conduct of the study or is an immediate family member of such an individual.

Participants with an Autoimmune Disease (Cohort 9 Only)

For participants with an autoimmune disease, the exclusion criteria for healthy participants listed above apply, with the following additions:

1. Concurrent use of the following medications/treatments:

* Systemic immunosuppressants/immunomodulators or other systemic treatments for autoimmune disease within 28 days or 5 half-lives (whichever is longer) before Day -1.
* Systemic antivirals or antifungals within 28 days prior to Day -1, or systemic antibiotics within 28 days prior to Day -1.
* Oral analgesics including opioids within 14 days prior to Day -1, except for acetaminophen at doses of <=2 g/day for relief of autoimmune disease-associated pain.
* Prescription and OTC medications other than those used for the treatment of an autoimmune disease within 14 days or 5 half-lives (whichever is longer) before Day -1, except for hormonal contraceptives, thyroid replacement medications, and medications used for the treatment of hypertension, diabetes mellitus (but not metformin), or hyperlipidemia which are permitted provided the medication(s) and dosage (dose and frequency) have been stable for at least 6 weeks prior to Day -1. Note that participants with thyroid hormone deficiency, hypertension, diabetes mellitus, or hyperlipidemia may be included in Part 3 of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) and Severity of AEs | Baseline up to Day 73
Part 1: Number of Participants who have Dose-limiting Adverse Reactions | Baseline up to Day 73
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Vital Sign Parameter | Baseline up to Day 73
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Physical Examination Findings | Baseline up to Day 73
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Electrocardiograms (ECGs) Parameters | Baseline up to Day 73
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Baseline up to Day 73
Part 2 and 3: Number of Participants with Adverse Events (AEs) and Severity of AEs | Baseline up to Day 94
Part 2 and 3: Number of Participants who have Dose-limiting Adverse Reactions | Baseline up to Day 94
Part 2 and 3: Number of Participants with Clinically Significant Changes from Baseline in Vital Sign Parameter | Baseline up to Day 94
Part 2 and 3: Number of Participants with Clinically Significant Changes from Baseline in Physical Examination Findings | Baseline up to Day 94
Part 2 and 3: Number of Participants with Clinically Significant Changes from Baseline in ECGs Parameters | Baseline up to Day 94
Part 2 and 3: Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Baseline up to Day 94

SECONDARY OUTCOMES:
Part 1: Maximum Serum Concentration (Cmax) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Time to Reach Maximum Serum Concentration (Tmax) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Area Under the Serum Concentration-time Curve from Zero to Time of the Last Quantifiable Concentration (AUC0-t) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Area Under the Serum Concentration-time Curve from Zero to infinity (AUC0-inf) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Elimination Half-life (t½) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Apparent Total Serum Clearance (CL/F) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Apparent Volume of Distribution Associated with the Terminal Phase (Vd/F) of LAD191 | Pre-dose, 4 hours and 8 hours post-dose on Days 1, 2, 3, 4, 6, 8, 15, 22, 29, 43, 57 and 71
Part 1: Number of Participants with Positive Anti-drug Antibodies (ADA) and Titer of ADA of LAD191 | Pre-dose on Day 1; 24 hours post-dose on Days 15; 48 hours post-dose on Days 43 and 71
Part 2: Area Under the Serum Concentration-time Curve from Zero to Time of the Last Quantifiable Concentration (AUC0-t) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Area Under the Concentration-time Curve within a Dosing Interval (AUCτau) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Maximum Serum Concentration (Cmax) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Time to Reach Maximum Serum Concentration (Tmax) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Minimum Serum Concentrations (Cmin) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Time to Cmin (tmin) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Area Under the Serum Concentration-time Curve from Zero to Time of the Last Quantifiable Concentration (AUC0-t) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Area Under the Concentration-time Curve within a Dosing Interval (AUCτau) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Maximum Serum Concentration (Cmax) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Time to Reach Maximum Serum Concentration (Tmax) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Minimum Serum Concentrations (Cmin) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Time to Cmin (tmin) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Apparent Total Serum Clearance (CL/F) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Apparent Volume of Distribution Associated with the Terminal Phase (Vd/F) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Elimination Half-life (t½) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2: Accumulation Ratios Based on AUC (R[AUC]) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours, 24 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 2 and 3: Number of Participants with Positive ADA and Titer of ADA of LAD191 | Pre-dose on Days 1, 15, and 29; 4 hours post-dose on Days 43; 48 hours post-dose on 64 and 92
Part 3: Area Under the Serum Concentration-time Curve from Zero to Time of the Last Quantifiable Concentration (AUC0-t) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Area Under the Concentration-time Curve within a Dosing Interval (AUCτau) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Maximum Serum Concentration (Cmax) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Time to Reach Maximum Serum Concentration (Tmax) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Minimum Serum Concentrations (Cmin) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Time to Cmin (tmin) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Area Under the Serum Concentration-time Curve from Zero to Time of the Last Quantifiable Concentration (AUC0-t) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Area Under the Concentration-time Curve within a Dosing Interval (AUCτau) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Maximum Serum Concentration (Cmax) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Time to Reach Maximum Serum Concentration (Tmax) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Minimum Serum Concentrations (Cmin) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Time to Cmin (tmin) at Steady State of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Apparent Total Serum Clearance (CL/F) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Apparent Volume of Distribution Associated with the Terminal Phase (Vd/F) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Elimination Half-life (t½) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92
Part 3: Accumulation Ratios Based on AUC (R[AUC]) of LAD191 | Pre-dose at Days 1, 8, 15, 22, 29, and 36; At 4 hours and 48 hours post-dose on Days 1, 36, 40, 43, 50, 64, 85 and 92

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (3):
- United States (3):
  - Doral Medical Research, Miami, Florida
  - Jennifer Parish, MD, Philadelphia, Pennsylvania
  - ICON Early Phase Services, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No